CLINICAL TRIAL: NCT04160871
Title: Efficacy of "Family Connections", a Program for Relatives of People With Borderline Personality Disorder in Spanish Population: A Study Protocol for a Randomized Control Trial
Brief Title: "Family Connections": a Program for Relatives of People With Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJaumeI19-1
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Relatives
Keywords: borderline personality disorder; family connections; relatives; dbt; intervention; program; caregivers
MeSH Terms: conditions — Borderline Personality Disorder; Maple syrup urine disease, type 2 | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized, Efficacy Study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Connections (Experimental): Experimental group
  Interventions: Behavioral: Family Connections
- Treatment As Usual (Active Comparator): Control group
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Family Connections — Intervention includes 12 sessions that follow a group format of 2 hours with a weekly frequency. FC program (Hoffman and Fruzzetti, 2005) is divided into six modules: 1: Updated information and research on BPD; 2: Psychoeducation on the development of BPD, available treatments and comorbidity; 3: Individual skills: self-control of emotions, mindfulness, reality acceptance skills, validation skills, etc. and skills of relationship to promote emotional well-being problem management (family skills); 4: Family skills to improve the quality of relationships in family interactions; 5: Communication skills and effective self-expression; and 6: Problem management. All modules include Practice exercises and homework. In addition, throughout the program, in order to increase social support, the FC program provides a forum where participants can stay in touch, share common problems and solutions.
  Arms: Family Connections
Behavioral: Treatment As Usual — The intervention lasts for 3 months and includes 12 sessions that follow a group format of 2 hours and with a weekly frequency. It includes the following components: Psychoeducation about personality disorders and, specifically, BPD and how these disorders evolve. Problems associated with BPD (eg, alcohol and / or drug use, eating disorders, etc.). The importance of "modeling" in family members: change of attitude towards difficult situations to reduce the escalation of tension and re-establish a healthy relationship between the patient and family. The handling of problems. Crisis management: Development of safe plans for when the patient is in emotional escalation.
  Arms: Treatment As Usual

SUMMARY:
The aim of this study is to validate an intervention for relatives of people with borderline personality disorder in Spanish population in a randomized control trial.

DETAILED DESCRIPTION:
Family members of patients with borderline personality disorder (BPD) often experience high levels of suffering, anxiety, stress, burden and helplessness. The treatment program with the most empirical support is "Family Connections". It is one of the first programs specifically designed to help relatives of patients with BPD. The program is an adaptation of multiple strategies of Dialectical Behavioral Therapy. It consists of 12 sessions with an approximate duration of two hours each. The results of these studies and their subsequent replications showed an improvement in family attitudes and perceived burden. The investigators have translated and adapted the program so that it could be applied to the Spanish population. The aim of the present study is to evaluate the effectiveness of the adaptation of "Family connections" in Spanish population through a controlled clinical trial. The first hypothesis of the study is that "Family Connections" will be more effective (significant reduction in the primary outcome variables), compared with a Treatment As Usual (TAU), in the posttest time and in the follow-ups of 3 and 6 months. In addition, a second hypothesis is that "Family Connections" will be more efficient (fewer abandonments, better opinion on the part of the patients) than TAU.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Having a relative with DSM-5 diagnosis of Personality Disorder
* Understand spoken and written Spanish.
* Grant informed consent.

Exclusion Criteria:

* Diagnosis of severe mental disorder.
* Presence of medical illness that may interfere with psychological treatment.
* Suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Burden Assessment Scale (BAS; Reinhard & Horwitz, 1992). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Burden Assessment Scale (BAS) consists of 19 items and it assess the caregivers' objective and subjective burden within the past six months. Items are rated on a 4-point Likert scale ranging from 1(nothing) to 4 (a lot), and higher values indicate stronger burden. Internal reliability of the scale ranged from .89 to .91 and it shows adequated validity (Reinhard, Gubman, Horwitz & Minsky, 1994).
Family Assessment Device - Global Functioning Scale (FAD-GFS; Epstein, Baldwin & Bishop, 1983). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Family Assessment Device - Global Functioning Scale (FAD-GFS) is a self-report questionnaire (Epstein, Baldwin & Bishop, 1983). It consists of 60 items about family functioning. It is composed of seven subscales: Problem-Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behavior Control and General Functioning. Items are rated on a 4-point Likert scale ranging from 1 (totally agree) to 4 (totally disagree), and higher scores indicate unhealthy functioning. Cronbach's alphas ranges from .72 to .83 for the subscales and general functioning is .92 (Miller, Epstein, Bishop & Keitner, 1985) and test-retest for the FAD scales were adequate (Miller, Epstein, Bishop & Keitner, 1985).

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21; Lovibond & Lovibond, 1995). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Depression, Anxiety and Stress Scale (DASS) have 42 items about negative emotional symptoms (Lovibond & Lovibond, 1995). Lovibond & Lovinbod (1995) proposed that a part of these subscales for can become part of a short version creating a new questionnaire of 21 items. Items are rated on a 4-point Likert scale ranging from 0 (It did not happen to me) to 3 (It happened to me a lot or most of the time), and higher scores indicate worse symptoms of depression, anxiety or stress. DASS-21 showed fantastic factor structures. Regarding to the internal consistency, Cronbach's alphas were excellent for the DASS-21 subscales: Depression (α = .94), Anxiety (α = .87) and Stress (α = .91) (Antony, Bieling, Cox, Enns & Swinson, 1998).
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004; Hervás & Jódar, 2008). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  We used the spanish version of the instrument Difficulties in Emotion Regulation Scale (DERS), developed by Gratz y Roemer (2004), with the aim to assess the emotional regulation problem. The scale was adapted to spanish and it was reduced from 36 items to 28 items (Hervás & Jódar, 2008). In this version, they figured on 5 scales instead 6 considering that "difficulties in the impulse control" and "limited access to regulation strategies" were joined into one named "emotional lack of control". The subscales are life interference, emotional confusion, emotional rejection, emotional lack of control and lack of emotional attention. Items are rated on a 5-point Likert scale ranging from 1 (rarely) to 5 (almost always), and higher scores indicate greater impairment or dysregulation. The psychometric properties show high consistency were Cronbach's alphas of the subscales range from .73 to .91 and .93 for the total scale (Hervás & Jódar, 2008).
Family Empowerment Scale (FES; Koren, DeChillo & Friesen, 1992). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Family Empowerment Scale (FES) consists of 34 items divided in three subscales: family, service system, and involvement in community that is refered to three ways of empowerment, attitudes, knowledge, and behaviors (Koren, DeChillo & Friesen, 1992). Items are rated on a scale of 1 (completely false) to 5 (totally true), and higher scores indicate a greater sense of empowerment. The psychometric properties are the following: regarding to the internal consistency of FES subscores, the coefficients ranged from .87 to .88 and validity and reliability are adequated (Koren, DeChillo & Friesen, 1992).
Connor-Davidson Resilience Scale (CD-RISC; Connor & Davidson, 2003). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Connor-Davidson Resilience scale is a 25-item measure of resilience. Items are rated on a 5-point Likert scale ranging from 0 (absolutely not) to 4 (almost always) and the punctuation is based on how the participant has felt over the last month. Higher scores means greater resilience (Connor & Davidson, 2003). The CD-RISC authors reported acceptable test-retest reliability (r = 0.87) and strong internal consistency (α = .89) (Connor & Davidson, 2003).
Quality of Life Index-Spanish Version (QLI-Sp; Mezzich, Cohen, Ruipérez & Yoon, 1999). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Quality of Life Index-Spanish Version consist of 10 items that assess aspects as physical, psychological/emotional well-being, self-care and independent functioning, occupational and interpersonal functioning, social-emotional and community and services support, personal and spiritual fulfillment and global perception of quality life. Items are rated on a scale of 1 (bad) to 10 (excellent), and higher scores means higher quality of life. This instrument has good psychometric properties as Cronbach's alpha of .89 and high test-retest reliability (r = 0.87) (Mezzich et al., 2000).
Beck Hopelessness Scale (BHS; Beck, Weissman, Lester & Trexler, 1974). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Beck Hopelessness Scale is a 20-item true-false instrument utilized for the measurement of hopelessness. It evaluates the attitude of the participant in the previous week. Nine items assess attitudes about the future and eleven items assess pessimistic statements. Items are rated as true or false, and higher scores reflects higher levels of hopelessness. Good psychometric properties are shown in this instrument. Internal consistency was excellent (α = .93) (Beck, Weissman, Lester & Trexler, 1974).
Openness To the Future Scale (OFS; Botella et al., 2018). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Openness Towards the Future Scale is a 10-items self-report that measures positive affective orientation towards the future. Items are rated on a 5-point Likert scale ranging from 1 (totally disagree) to 5 (totally agree), and higher scores indicate better openness to the future. It shows adequate psychometric properties for both clinical and general samples. Cronbach's alpha was acceptable for both clinical (α = .82) and community samples (α = .87) (Botella et al., 2018).
Personality Inventory for DSM-5 (PID-5; Krueger, Derringer, Markon, Watson & Skodol, 2012). | Pre-treatment
  Personality Inventory for DSM-5 (PID-5) is a 220-item instrument that assesses 25 traits, which form five domains (Negative Affectivity, Detachment, Antagonism, Disinhibition, and Psychoticism). The 25 traits are the following: Anhedonia, Anxiousness, Attention Seeking, Callousness, Deceitfulness, Depressivity, Distractibility, Eccentricity, Emotional Lability, Grandiosity, Hostility, Impulsivity, Intimacy Avoidance, Irresponsibility, Manipulativeness, Perceptual Dysregulation, Perseveration, Restricted Affectivity, Rigid Perfectionism, Risk Taking, Separation Insecurity, Submissiveness, Suspiciousness, Unusual Beliefs and Experiences, and Withdrawal. Items are ranged on a 4-point Likert scale ranging from 0 (totally disagree) to 3 (totally agree), and higher average scores indicate more "dysfunction" in a specific personality trait facet or domain. Internal consistency ranged from .72 to .96 with a median of .86 (Krueger, Derringer, Markon, Watson & Skodol, 2012).
Structured Clinical Interview for DSM-IV Axis II (SCID-II; First, Gibbon, Spitzer, Williams & Benjamin, 1997). | Pre-treatment
  Structured Clinical Interview for DSM-IV Axis II consists of a semistructured format involving 10 standard DSM-IV personality disorders and the Personality Disorder Not Otherwise Specified, Depressive Personality Disorder and Passive-Aggressive Personality Disorder. Items are rated as "yes" or "no", and two or more scores on "yes" mean that participant may have a personality disorder and should be evaluated with the interview, and you have to assess the personality disorder depending on the punctuation of each (5 items or more: dependent, depressive, squizotypal, histrionic, narcissistic and borderline; 4 items or more: avoidant, obsessive-compulssive, passive-agressive, paranoid and schizoid; 3 items or more: antisocial; 1 item or more: non-specified. Adequate inter-rater reliability coefficients were reported (.48-.98) and satisfactory internal consistency coefficients (ranges from .71 to .94) (Maffei et al. 1997).

OTHER OUTCOMES:
Family Assessment Device - Global Functioning Scale (FAD-GFS; Epstein, Baldwin & Bishop, 1983). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  This instrument is also carried out in the evaluation of patients. Family Assessment Device - Global Functioning Scale (FAD-GFS) is a self-report questionnaire (Epstein, Baldwin & Bishop, 1983). It consists of 60 items about family functioning. It is composed of seven subscales: Problem-Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behavior Control and General Functioning. Items are rated on a 4-point Likert scale ranging from 1 (totally agree) to 4 (totally disagree), and higher scores indicate unhealthy functioning. Cronbach's alphas ranges from .72 to .83 for the subscales and general functioning is .92 (Miller, Epstein, Bishop & Keitner, 1985) and test-retest for the FAD scales were adequate (Miller, Epstein, Bishop & Keitner, 1985).
Depression, Anxiety and Stress Scale (DASS-21; Lovibond & Lovibond, 1995). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  This instrument is also carried out in the evaluation of patients. Depression, Anxiety and Stress Scale (DASS) have 42 items about negative emotional symptoms (Lovibond & Lovibond, 1995). Lovibond & Lovinbod (1995) proposed that a part of these subscales for can become part of a short version creating a new questionnaire of 21 items. Items are rated on a 4-point Likert scale ranging from 0 (It did not happen to me) to 3 (It happened to me a lot or most of the time), and higher scores indicate worse symptoms of depression, anxiety or stress. DASS-21 showed fantastic factor structures. Regarding to the internal consistency, Cronbach's alphas were excellent for the DASS-21 subscales: Depression (α = .94), Anxiety (α = .87) and Stress (α = .91) (Antony, Bieling, Cox, Enns & Swinson, 1998).
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004; Hervás & Jódar, 2008). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  This instrument is also carried out in the evaluation of patients. Difficulties in Emotion Regulation Scale (DERS), developed by Gratz y Roemer (2004), with the aim to assess the emotional regulation problem. The scale was adapted to spanish and it was reduced from 36 items to 28 items (Hervás & Jódar, 2008). In this version, they figured on 5 scales instead 6 considering that "difficulties in the impulse control" and "limited access to regulation strategies" were joined into one named "emotional lack of control". The subscales are life interference, emotional confusion, emotional rejection, emotional lack of control and lack of emotional attention. Items are rated on a 5-point Likert scale ranging from 1 (rarely) to 5 (almost always), and higher scores indicate greater impairment or dysregulation. The psychometric properties show high consistency were Cronbach's alphas of the subscales range from .73 to .91 and .93 for the total scale (Hervás & Jódar, 2008).
Lum Emotional Availability of Parents (LEAP; Lum & Phares, 2005). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Lum Emotional Availability of Parents consists of 15 items that involves participants' mothers and fathers emotional availability. Items are rated on a 6-point Likert scale ranging from 1 (never) to 6 (always), and higher scores indicate better emotional availability. Internal consistency was excellent for non-clinical sample for the mother form (α = .96) and for father form (α = .97); also for the mother form in a clinical sample (α = .92), and for the father form (α = .93). This instrument has adequated test-retest reliability for the mother form (r = .92) and for the father form (r = .85) (Lum & Phares, 2005).
Validating and Invalidating Responses Scale (VIRS; Fruzzetti, 2007). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month-follow-up.
  Validating and Invalidating Responses Scale is a 16-items self-report which evaluates levels of validation and invalidation of caregiver's responses. This instrument has two subscales: validation and invalidation responses. This two are moderately correlated. Items are rated on a 5-point Likert scale, ranging from 0 (never) to 4 (almost all the time), and higher scores indicate more perceived validation or invalidation from the caregiver who is assessed. There are no psychometric properties available on the VIRS yet.
Post-Module measures (P-M) | Immediately after the intervention
  Post-Module is an instrument constructed by our research team oriented to assess the level of change obtained with respect to the therapeutic modules as well as the degree of satisfaction to receive the treatment. It evaluates the six modules of the treatment in the two conditions. There are two subscales: one evaluates the learning of the abilities of the module and it is rated from 0 (nothing) to 10 (a lot), and the other evaluates how the module has helped to the caregiver to improve several aspects such as knowing and understanding the problem, emotion's comprehension, mindfulness of the relationship with their relative, acceptance, family atmosphere and problem solving on the family atmosphere, and it is rated from 1 (nothing) to 4 (a lot). Expectation scale is assessed on the end of the first module.

CONTACTS AND LOCATIONS:
Overall Officials: José Heliodoro Marco Salvador, Dr, Principal Investigator — University of Valencia; Isabel Fernández Felipe, PhD student, Principal Investigator — Universitat Jaume I; Amanda Díaz García, Dr, Principal Investigator — Universitat Jaume I; Cristina Botella Arbona, Dr, Principal Investigator — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication.
Access Criteria: The data will be available to anyone who wishes to access them.

REFERENCES:
- [Background] Hoffman PD, Fruzzetti AE. Advances in interventions for families with a relative with a personality disorder diagnosis. Curr Psychiatry Rep. 2007 Feb;9(1):68-73. doi: 10.1007/s11920-007-0012-z. PMID 17257517
- [Background] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Background] Hoffman PD, Buteau E, Hooley JM, Fruzzetti AE, Bruce ML. Family members' knowledge about borderline personality disorder: correspondence with their levels of depression, burden, distress, and expressed emotion. Fam Process. 2003 Winter;42(4):469-78. doi: 10.1111/j.1545-5300.2003.00469.x. PMID 14979218
- [Background] Hoffman PD, Fruzzetti AE, Swenson CR. Dialectical behavior therapy--family skills training. Fam Process. 1999 Winter;38(4):399-414. doi: 10.1111/j.1545-5300.1999.00399.x. PMID 10668619
- [Background] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Background] Rajalin M, Wickholm-Pethrus L, Hursti T, Jokinen J. Dialectical behavior therapy-based skills training for family members of suicide attempters. Arch Suicide Res. 2009;13(3):257-63. doi: 10.1080/13811110903044401. PMID 19590999
- [Derived] Guillen V, Bolo S, Fonseca-Baeza S, Perez S, Garcia-Alandete J, Botella C, Marco JH. Psychological assessment of parents of people diagnosed with borderline personality disorder and comparison with parents of people without psychological disorders. Front Psychol. 2023 Jan 13;13:1097959. doi: 10.3389/fpsyg.2022.1097959. eCollection 2022. PMID 36710828
- [Derived] Fernandez-Felipe I, Guillen V, Marco H, Diaz-Garcia A, Botella C, Jorquera M, Banos R, Garcia-Palacios A. Efficacy of "Family Connections", a program for relatives of people with borderline personality disorder, in the Spanish population: study protocol for a randomized controlled trial. BMC Psychiatry. 2020 Jun 15;20(1):302. doi: 10.1186/s12888-020-02708-8. PMID 32539740